CLINICAL TRIAL: NCT01564615
Title: Reduction of Catheter-Related Bloodstream Infections in Preterm Infants by the Use of Catheters With the AgION Antimicrobial System
Brief Title: AgION Catheter for Preventing Catheter-Related Bloodstream Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Dani, Associate Professor of Pediatrics, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01/2012
Record Dates: First submitted 2012-03-19; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Catheter-Related Infections
Keywords: Catheter related bloodstream infection; Umbilical venous catheter; Silver; Preterm infants
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AgION catheter (Experimental): Patients in this arm received an AgION impregnated catheter (4.0-5.0 F Lifecath PICC ExpertTM, Vygon, Ecouen, France).
  Interventions: Device: Umbilical catheterization (AgION )
- Non-impregnated polyurethane catheter (Active Comparator): Patients in this arm received a non-impregnated polyurethane umbilical catheter (3.5-5.0 F ArgyleTM, Kendall, Tullamore, Iceland)
  Interventions: Device: Umbilical catheterization (ArgyleTM)

INTERVENTIONS:
Device: Umbilical catheterization (AgION ) — Infants received a AgION impregnated catheter (4.0-5.0 F Lifecath PICC ExpertTM, Vygon, Ecouen, France).
  Arms: AgION catheter
Device: Umbilical catheterization (ArgyleTM) — Infants received a polyurethane non-impregnated catheter (3.5-5.0 F ArgyleTM, Kendall, Tullamore, Iceland)
  Arms: Non-impregnated polyurethane catheter

SUMMARY:
The investigators assessed if use of AgION-impregnated umbilical catheters can decrease the occurrence of catheter-related bloodstream infections (CRBSI) in preterm infants.

DETAILED DESCRIPTION:
Recently, a silver zeolite-impregnated catheter has been commercialized. This material, namely the patented silver compound AgION™, releases antimicrobially active silver ions which may help prevent catheter-related bloodstream infections CRBSIs which are frequent in preterm infant.

The investigators hypothesized that the use of AgION-impregnated umbilical catheters could decrease the occurrence of CRBSIs in preterm infants. To assess this hypothesis the investigators carried out a randomized controlled study in which preterm infants needing an umbilical vein catheter would received either an AgION catheter or a traditional non-impregnated polyurethane catheter.

Infants with gestational age < 30 weeks were randomized to receive an AgION- impregnated or non-impregnated polyurethane umbilical venous catheter (UVC) by opening sealed opaque envelopes. The primary end point was the incidence of CRBSIs during the time the UVC was in place.

The investigators studied 86 infants, 41 of whom received the AgION catheter and 45 the non-impregnated catheter. During umbilical venous catheterization 2% of infants in the AgION group developed CRBSI in comparison with 22% of infants in the control group (p=0.005). The incidence density of CRBSIs during the study period was lower in infants who received AgION catheters compared to the control group (2.1/1000 catheter days versus 25.8/1000 catheter days; p<0.001). The occurrence of UVC colonization was similar in both groups. The Kaplan-Meier estimates of the cumulative likelihood of being free of a CRBSI at each day of UVC placement demonstrate the statistically significant (p=0.004) protective effect of AgION impregnated catheters. Moreover, infants in the AgION group had shorter hospital stay (p=0.04), and a lower case fatality rate due to BSI (p=0.01) than infants in the control group.

AgION catheters were well tolerated and none of patients showed signs attributable to silver toxicity.

Multivariate analysis demonstrated that non-impregnated catheter use (OR 12.5, 95% C.l. 2.06-75.9) and catheter placement for more than 7 days (OR 5.1, 95% C.l. 1.13-23.6) increased the risk of developing a CRBSI in our population.

Conclusions. The AgION-impregnated UVCs were effective in decreasing the development of CRBSIs in preterm infants compared to non-impregnated polyurethane UVCs.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 30 weeks
* Need of an umbilical venous catheter in the first week of life
* Parental informed consent.

Exclusion Criteria:

* Major congenital malformations
* Hydrops fetalis
* Inherited congenital metabolic diseases
* Death during the first week of life

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Incidence of CRBSIs | Infants were followed for the duration the AgION umbilical venous catheter (UVC) was in place, an expected average of 10 days
  We evaluated the incidence of CRBSIs (definite plus probable) during the time the UVC was in place.

SECONDARY OUTCOMES:
Infection density | Infants were followed for the duration the AgION umbilical venous catheter (UVC) was in place, an expected average of 10 days
  Number of infections/1000 catheter days, likelihood of freedom from CRIBSIS, and signs of catheter intolerance and possible adverse effects from silver ion toxicity were evaluated for the duration of umbilical venous catheterization; occurrence of BPD, IVH, PVL, ROP, and NEC, length of stay in hospital, case fatality rate for infants with CRBSI, and death were evaluated at discharge.
Likelihood of freedom from CRIBSIs | Infants were followed for the duration the AgION umbilical venous catheter (UVC) was in place, an expected average of 10 days
  Likelihood of freedom from CRIBSIS for the duration of umbilical venous catheterization
AgION catheters tolerability | Infants were followed for the duration the AgION umbilical venous catheter (UVC) was in place, an expected average of 10 days
  Signs of local intolerance, such as skin infection, were recorded. We also evaluated possible adverse effects from silver ion toxicity, such as the occurrence of argyria (blue-grey discoloration of the skin) or hepatic damage (i.e.: increase in AST/ALT enzymes).
Case fatality rate for infants with CRBSI | Hospital stay duration, an expected average of 80 days
  We evaluated the mortality caused by CRBSI in infants who received AgION-impregnated and non-impregnated groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Dani, MD, Principal Investigator — Department of Surgical and Medical Critical Care, Section of Neonatology, University of Florence
Locations (1):
- Careggi Univesity Hospital, Florence, Italy, Italy